CLINICAL TRIAL: NCT01311531
Title: Treatment of Distal Radial Fractures With Volar Locking Plates Versus Fragment-specific Fixation (TriMed Classic). A Randomized Trial
Brief Title: Volar Locking Plate vs Fragment Specific Fixation in Wrist Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETIK 2009/318
Record Dates: First submitted 2011-03-03; First posted 2011-03-09 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Distal Radius Fractures
Keywords: Fracture; Radius; Surgery; Osteosynthesis
MeSH Terms: conditions — Wrist Fractures; Fractures, Bone | interventions — Open Fracture Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TriMed fragment-specific fixation (Active Comparator)
  Interventions: Procedure: Open reduction and fixation with TriMed fragment-specific system
- TriMed volar locking plate (Active Comparator)
  Interventions: Procedure: Open reduction and fixation with TriMed volar locking plate

INTERVENTIONS:
Procedure: Open reduction and fixation with TriMed fragment-specific system — Anatomical reduction, achieved by the open technique.
  Arms: TriMed fragment-specific fixation
Procedure: Open reduction and fixation with TriMed volar locking plate — Anatomical reduction, achieved by the open technique.
  Arms: TriMed volar locking plate

SUMMARY:
The treatment of unstable, non-reducible distal radial fractures is still controversial. The aim of the present study is to compare the subjective, clinical and radiographic outcome of the TriMed fragment-specific system with a volar locking plate in patients with unstable, non-reducible and also redislocated distal radial fractures.

DETAILED DESCRIPTION:
The distal radial fracture is one of the most common fractures, with an annual incidence in southern Sweden of 26 per 10,000 inhabitants (Brogren et al. 2007). Non-surgical treatment, predominantly plaster cast or simple splints, comprises the basic treatment in non-displaced fractures, as well as in displaced, but reducible fractures (Handoll and Madhok 2003). In the unstable, non-reducible distal radial fractures, surgical treatment is necessary but can be complex. The choice of method is still controversial (Chen and Jupiter 2007), especially regarding the result over time (Downing and Karantana 2008). External fixation has been the preferred method of operation for decades, but with the introduction of the volar locking plate technique, internal fixation has rapidly become more and more popular, without any solid foundation in the evidence-based medicine (Margaliot et al. 2005).

We have shown in a randomized study that open reduction and internal fixation of distal radial fractures using the TriMed fragment-specific system resulted in better grip strength and forearm rotation at 1-year follow up than closed reduction and bridging external fixation (Abramo et al. 2009). Later we followed up the same cohort at a mean of 5-years, with the primary aim of determining whether the superior results of internal fixation in unstable distal radial fractures persist over time. The conclusion of this study was that, internal fixation is better than external fixation regarding grip strength and forearm rotation at 1-year but the difference disappears at the 5-year follow-up as both groups approach normal values (Landgren et al. submitted in 2010).

The aim of the present study is to compare the subjective, clinical and radiographic outcome of the TriMed fragment-specific system with a volar locking plate in patients with unstable, non-reducible and also redislocated distal radial fractures. The patients who meet all eligibility criteria and provide consent to participate will be randomly assigned to reduction and fixation with either volar locking plate or Trimed fragment-specific system. Patients will undergo physiotherapy, clinical evaluation, radiographic evaluation at fixed intervals and will also include QuickDASH, VAS, SF-12 and EQ5D. There will be 25 patients in each arm and the patients will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* AO type A or C fracture, unstable and non-reducible at day of trauma.
* AO type A or C fracture, redislocated at the 14 day clinical and radiological control.
* Incongruent RC-joint or DRU-joint and/or axial compression > 2 mm and/or dorsal compression 20°.

Exclusion Criteria:

* Previous fracture of the same wrist
* Volar Barton fractures (AO Type B)
* Fracture on the other side or other concomitant fracture that also needs treatment.
* Open fracture
* Fracture expansion to the diaphysis
* Ongoing chemo- or radiotherapy
* Metabolic diseases that affect the bone
* Dementia, mental illness, alcohol abuse or difficulty understanding the language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Grip strength | 12 months
  Will be measured by a physiotherapist at 6 weeks, 3 months and 12 months. Evaluated at 12 months.

SECONDARY OUTCOMES:
Forearm rotation (pronation/supination) measured in degrees | 6 weeks, 3 months and 12 months
  The evaluation of ange forearm rotation or range of motion preformed by a physiotherapist. It will be measured in degrees with a goniometer.
Subjective outcome measured with QuickDASH (scale 0-100) | 0, 6 weeks, 3 and 12 months
  The patients own evaluation of their arm will be measured using the QuickDASH (Quick Disabilities of the Arm Shoulder and Hand).
Visual Analog Scale | 0, 6 weeks, 3 and 12 months
  The Visual Analog Scale (VAS) will be used to evaluated different parameters: pain in rest, pain in work, function and cosmetic appearance of the hand
Number of reoperations | 12 months
  Number of participants with adverse events as a measure of safety and tolerability will be preformed
EQ-5D | 0, 6 weeks, 3 and 12 months
  The standardised EQ-5D instrument will be used as a measure of health outcome

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Tägil, MD, Principal Investigator — Department of Hand Surgery Malmö/Lund, Lund University and Skåne University Hospital, Lund, Sweden
Locations (1):
- Department of Hand Surgery Malmö/Lund, Lund University and Skåne University Hospital, Lund, Sweden, Lund, Sweden

REFERENCES:
- See also: Abramo et al. 2009 — http://www.ncbi.nlm.nih.gov/pubmed/19857180